CLINICAL TRIAL: NCT06770959
Title: Frequency of Gastrointestinal and Hepatic Manifestations Among Patients with Multiple Sclerosis, a Clinical Hospital Based Study
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Nayera Mohamed Refaat Abdelhameed, doctor, Assiut University
Other Study IDs: GIT symptoms in MS patients
Record Dates: First submitted 2024-12-27; First posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: MS (Multiple Sclerosis)
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The aim of this work is to identify different pattern of Gastrointestinal and Hepatic symptoms and its Frequency among patients with Multiple Sclerosis

DETAILED DESCRIPTION:
Historically, the routine evaluation of symptoms in MS patients focused on skeletal muscle impairments that restricted mobility. Within the last two decades, symptoms such as dysphagia, bladder and bowel dysfunction, among others, have been increasingly recognized and incorporated into patient assessments [1-3]. The GI problems felt to be most common in MS patients involve deglutition and defecation and require volitional muscle coordination. This association may link the development of such GI problems to underlying MS disease progression. However, GI symptoms that are not dependent upon skeletal muscle control are common in the general population and may also be present in MS patients. More than two decades ago, Hinds and colleagues described a high prevalence of anorectal dysfunction in a large cohort of MS patients [4]. Since then, the diagnostic and clinical approach to MS care has changed dramatically and now emphasizes the early introduction of disease modifying therapies [5]. However, despite changes in MS care, anorectal dysfunction and swallowing problems continue to be an important problem for MS patients . Little is known about other GI symptoms in MS patients in this new era of pervasive use of disease modifying therapies. To address this gap in knowledge, the investigators sought to define the prevalence of GI symptoms and syndromes in a large sample of contemporary MS patients

ELIGIBILITY:
Inclusion Criteria:

* 1- both sex 2- All patients diagnosed MS ( in recovery on DMT) according to the 2017-McDonalds criteria.

  3- Pt with MS suffer from git and hepatic symptoms not explained by known cause as Hepatitis virus،metabolic disorders as Wilson . hemochromatosis,etc Drug induced , Alcohol , Git symptoms as dysphagia, vomiting,reflux

  4- An informed consent will be obtained from all the patients, the study will be approved by ethical committee in faculty of Medicine Assiut University

Exclusion Criteria :1-patients already diagnosed with other GIT disorders before diagnosis of MS

2_ Presence of other disorder or on medications that may affect the neurological or GIT disorders.

3_ Patients failed to commit to the follow up visits and regular MRI scans 4_ Patients refused to sign the written informed consent Patients who will meet the inclusion and exclusion criteria will be assessed in the 1st visit by direct interview followed by clinical examination and neuropsychological assessments. Baseline MRI scans will be obtained at the first visit

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: both genders people on remission any age
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Detection of Prevalence of git and hepatic manifestation in people with MS and its relations to MS treatment | 24 month

REFERENCES:
- [Background] Levinthal DJ, Rahman A, Nusrat S, O'Leary M, Heyman R, Bielefeldt K. Adding to the burden: gastrointestinal symptoms and syndromes in multiple sclerosis. Mult Scler Int. 2013;2013:319201. doi: 10.1155/2013/319201. Epub 2013 Sep 17. PMID 24163768